CLINICAL TRIAL: NCT03362502
Title: A PHASE 1B MULTICENTER, OPEN-LABEL, SINGLE ASCENDING DOSE STUDY TO EVALUATE THE SAFETY AND TOLERABILITY OF PF-06939926 IN AMBULATORY AND NON-AMBULATORY SUBJECTS WITH DUCHENNE MUSCULAR DYSTROPHY
Brief Title: A Study to Evaluate the Safety and Tolerability of PF-06939926 Gene Therapy in Duchenne Muscular Dystrophy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: All participants who have received fordadistrogene movaparvovec in any Pfizer study will now be assessed for long-term safety in 1 combined study: C3391003
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C3391001; NCT03362502 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: gene therapy; mini-dystrophin; AAV; fordadistrogene movaparvovec
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PF-06939926 (Experimental)
  Interventions: Genetic: PF-06939926

INTERVENTIONS:
Genetic: PF-06939926 — Recombinant adeno-associated virus, serotype 9 (AAV9) carrying a truncated human dystrophin gene (mini-dystrophin) under the control of a muscle-specific promoter.
  Subjects will receive a single intravenous infusion of one of 2 dose levels.

SUMMARY:
This is a first-in-human/first-in-patient, multi-center, open-label, non-randomized, ascending dose, safety and tolerability study of a single intravenous infusion of PF-06939926 in ambulatory and non-ambulatory subjects with Duchenne muscular dystrophy (DMD). Other objectives include measurement of dystrophin expression and distribution, and assessments of muscle strength, quality, and function.

A total of approximately 22 subjects will receive PF-06939926, and these will include both ambulatory and non-ambulatory subjects. Up to 13 subjects may be included in a cohort that includes the concomitant medication, sirolimus. In order to mitigate unanticipated risks to subject safety, enrollment will be staggered within and between two planned dose-levels and will include a formal review by an external data monitoring committee (E-DMC) prior to dose progression.

ELIGIBILITY:
Inclusion Criteria:

* Age as follows, based on ambulatory status:

  * FOR AMBULATORY PARTICIPANTS, defined as the ability to walk at least 10 meters unassisted: Between 4 and 12 years, inclusive,
  * FOR NON-AMBULATORY PARTICIPANTS, defined as the inability to walk at least 10 meters unassisted: No age restrictions so long as loss of ambulation occurs prior to the subject's 17th birthday;
* Diagnosis of Duchenne muscular dystrophy confirmed by medical history and genetic testing;
* Receipt of glucocorticoids for 6 months and a stable daily dose for at least 3 months prior to study entry;
* Ability to tolerate magnetic resonance imaging (MRI) without sedation and with no contraindications to these procedures;
* Ability to tolerate muscle biopsies under anesthesia with no contraindications to these procedures;
* Body weights as follows, based on ambulatory status:

  * FOR AMBULATORY PARTICIPANTS: Between 15 kg and 50 kg,
  * FOR NON-AMBULATORY PARTICIPANTS: Less than 75 kg, but which may be managed or adjusted to a lower limit, especially to ensure participant safety;
* Functional performance as follows, based on ambulatory status:

  * FOR AMBULATORY PARTICIPANTS: Ability to rise from floor within seven (7) seconds,
  * FOR NON-AMBULATORY PARTICIPANTS: Percent predicted forced vital capacity greater than 40% as part of pulmonary function tests, as well as adequate upper limb function.

Exclusion Criteria:

* Receipt of live attenuated vaccination within 3 months prior to receiving PF-06939926 or exposure to an influenza (or other inactivated) vaccination or systemic antiviral and/or interferon therapy within 30 days prior to receipt of PF-06939926;
* Prior exposure to any gene therapy agent, including exon-skipping agents;
* Exposure to other investigational drugs within 30 days or 5 half-lives, whichever is longer;
* Neutralizing antibodies (NAb) against adeno-associated virus, serotype 9 (AAV9);
* Compromised cardiac function as indicated by left ventricular ejection fraction on cardiac MRI, as follows, based on ambulatory status:

  * FOR AMBULATORY PARTICIPANTS: Less than 55%,
  * FOR NON-AMBULATORY PARTICIPANTS: Less than 35%;
* Inadequate hepatic or renal function or risk factors for autoimmune disease on screening laboratory assessments.
* The following genetic abnormalities in the dystrophin gene as confirmed by the investigator based on the review of the DMD genetic testing:

  1. Any mutation (exon deletion, exon duplication, insertion, or point mutation) affecting any exon between exon 9 and exon 13, inclusive; OR
  2. A deletion that affects both exon 29 and exon 30.

Sirolimus Cohort

Inclusion Criteria

* > 8 years of age Exclusion Criteria
* Hypersensitivity to sirolimus or intolerance to soy, including a history of angioedema
* Concomitant use with strong CYP3A4/P-gp inducers or inhibitors

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2025-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - MRI Research Center, Los Angeles, California
  - Reed Neurological Research Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Investigational Drug Section), Los Angeles, California
  - Ronald Reagan UCLA Medical Center - Interventional Radiology, Los Angeles, California
  - Ronald Reagan UCLA Medical Center Drug Information Center, Los Angeles, California
  - UCLA (David Geffen School of Medicine), Los Angeles, California
  - UCLA Children's Heart Center, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UCLA Outpatient Surgery Center, Los Angeles, California
  - Duke Neurology, Durham, North Carolina
  - Duke University Medical Center, Lenox Baker Children's Hospital, Durham, North Carolina
  - Biospecimen Repository & Processing Core - BPRC, Durham, North Carolina
  - Duke Cardiovascular Magnetic Resonance Center, Durham, North Carolina
  - Duke Children's Hospital & Health Center, Durham, North Carolina
  - Duke University Hospital Investigational Drug Services (IDS) Pharmacy, Durham, North Carolina
  - CCTS Clinical Research Center, Salt Lake City, Utah
  - University of Utah Imaging and Neurosciences Center, Salt Lake City, Utah
  - University of Utah Hospital & Clinics Investigational Drug Services, Salt Lake City, Utah
  - University of Utah Hospital, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Utah Clinical Neurosciences Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Walsh J, Palandra J, Duriga N, Beidler D, McIntosh A, Binks M, Neubert H. Dystrophin/mini-dystrophin expression analysis by immunoaffinity liquid chromatography-tandem mass spectrometry after gene therapy for DMD. Gene Ther. 2025 Dec;32(6):573-580. doi: 10.1038/s41434-025-00554-5. Epub 2025 Aug 2. PMID 40753271
- [Derived] Byrne BJ, Butterfield RJ, Shieh PB, Smith EC, Licht C, Binks M, Casinghino S, Delnomdedieu M, Ravindra KC, McDonnell T, Ryan K, Schulz M, Shen Q, Shi H, Sirivelu MP, Vaidya VS, Whiteley L, Levy DI. Complement activation in a phase Ib study of fordadistrogene movaparvovec for Duchenne muscular dystrophy. Mol Ther. 2025 Sep 3;33(9):4226-4238. doi: 10.1016/j.ymthe.2025.06.032. Epub 2025 Jun 28. PMID 40583275
- [Derived] Sherlock SP, Levy DI, McIntosh A, Shieh PB, Smith EC, McDonnell TG, Ryan KA, Delnomdedieu M, Binks M, Lal AK, Butterfield RJ. Cardiac safety of fordadistrogene movaparvovec gene therapy in Duchenne muscular dystrophy: Initial observations from a phase 1b trial. Mol Ther. 2025 Sep 3;33(9):4216-4225. doi: 10.1016/j.ymthe.2025.06.031. Epub 2025 Jun 28. PMID 40583273
- [Derived] Butterfield RJ, Shieh PB, Li H, Binks M, McDonnell TG, Ryan KA, Delnomdedieu M, Belluscio BA, Neelakantan S, Levy DI, Schwartz PF, Smith EC. AAV mini-dystrophin gene therapy for Duchenne muscular dystrophy: a phase 1b trial. Nat Med. 2025 Aug;31(8):2712-2721. doi: 10.1038/s41591-025-03750-3. Epub 2025 Jun 27. PMID 40579547
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3391001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study reached its primary completion date (PCD) on 28 Mar 2022. The data cutoff for PCD was on 30 Sep 2022. As of 30 Sep 2022, a total of 22 participants, including 19 ambulatory participants and 3 non-ambulatory participants, were enrolled and assigned to treatment.
Pre-assignment Details: One participant was enrolled but not dosed due to a pause in enrollment. The participant was considered as an early termination due to screening window running out. The participant was subsequently re-screened and assigned to study intervention with another participant ID. Therefore, a total of 22 unique participants were enrolled as of 30 Sep 2022.
Groups:
- PF-06939926: Low Dose, Ambulatory Cohort: Ambulatory participants received a single intravenous (IV) infusion of PF-06939926 1E+14 vector genomes per kilogram bodyweight (vg/kg) on Day 1, followed by at least 24 hours of in-patient monitoring, a 2-week follow-up visit, 1-year follow-up, and long-term follow-up for 4 years.
- PF-06939926: High Dose, Ambulatory Cohort: Ambulatory participants received a single IV infusion of PF-06939926 2E+14 vg/kg per transgene (TG)-based titer method or 3E+14 vg/kg per the inverted terminal repeats (ITR)-based titer method on Day 1, followed by at least 24 hours of in-patient monitoring, a 2-week follow-up visit, 1-year follow-up, and long-term follow-up for 4 years. PF-06939926 at 3E+14 vg/kg per the ITR-based titer method is approximately equivalent to 2E+14 vg/kg per the TG-titer method.
- PF-06939926: High Dose, Non-Ambulatory Cohort: Non-ambulatory participants received a single IV infusion of PF-06939926 2E+14 vg/kg per TG-based titer method or 3E+14 vg/kg per the ITR-based titer method on Day 1, followed by at least 24 hours of in-patient monitoring, a 2-week follow-up visit, 1-year follow-up, and long-term follow-up for 4 years. PF-06939926 at 3E+14 vg/kg per the ITR-based titer method is approximately equivalent to 2E+14 vg/kg per the TG-titer method.
Period: Overall Study
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Started | 3 | 16 | 3
Completed (Completed indicates participants completed the 1-year follow-up as of data cutoff on 30 Sep 2022.) | 3 | 16 | 2
Not Completed | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes all enrolled participants who received PF-06939926 as of the PCD data cutoff (30 Sep 2022). Participants were analyzed according to the intervention they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort | Total
Number analyzed (Participants) | 3 | 16 | 3 | 22
Age, Customized [Count of Participants; unit: Participants]
  6-<7 years | 0 | 2 | 0 | 2
  7-<8 years | 1 | 4 | 0 | 5
  8-<9 years | 1 | 4 | 0 | 5
  9-<10 years | 1 | 4 | 0 | 5
  10-<11 years | 0 | 1 | 0 | 1
  11-<12 years | 0 | 0 | 0 | 0
  >=12 years | 0 | 1 | 3 | 4
Age, Customized [Median (Full Range); unit: Years] | 8 [7 to 9] | 8 [6 to 12] | 14 [13 to 16] | 8 [6 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 16 | 3 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 13 | 1 | 17
  Black or African American | 0 | 1 | 1 | 2
  Asian | 0 | 2 | 0 | 2
  Not Reported | 0 | 0 | 1 | 1
Mutation Type [Count of Participants; unit: Participants] — Confirmation by genetic testing of the diagnosis of duchenne muscular dystrophy (DMD) was reported from an appropriate regulated laboratory using a clinically validated genetic test.
  Participants
    Deletion | 1 | 0 | 0 | 1
    Exon Deletion | 1 | 7 | 2 | 10
    Exon Duplication | 0 | 3 | 0 | 3
    Insertion | 0 | 1 | 0 | 1
    Point Mutation | 1 | 4 | 1 | 6
    Cryptic Splice Donor Site | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-Causality Treatment-Emergent Adverse Events (TEAEs) for 1-Year Follow-Up
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Any AE that started following start of treatment of PF-06939926 was counted as a treatment-emergent AE (TEAE). A serious AE (SAE) was an untoward medical occurrence that resulted in death, was life-threatening (immediate risk of death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect, or was considered to be an important medical event. Severe AE=an event that prevents normal everyday activities.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: Includes all enrolled participants who received PF-06939926. Participants were analyzed according to the intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  TEAEs | 3 | 16 | 3
  SAEs | 0 | 3 | 2
  Severe AEs | 1 | 2 | 2

2. Primary Outcome: Number of Participants With All-Causality TEAEs by System Organ Class (SOC) and Preferred Term (PT) for 1-Year Follow-Up
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Any AE that started following start of treatment of PF-06939926 was counted as a TEAE. For this outcome measure, TEAEs were reported according to Medical Dictionary for Regulatory Activities (MedDRA) version 25.0 SOC and PT.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, Total | 2 | 9 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Anaemia | 0 | 2 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Haemolysis | 0 | 1 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Haemolytic uraemic syndrome | 0 | 0 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Leukocytosis | 1 | 0 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Lymphopenia | 1 | 0 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Thrombocytopenia | 0 | 9 | 0
  SOC: CARDIAC DISORDERS, Total | 0 | 0 | 2
  SOC: CARDIAC DISORDERS, PT: Cardiogenic shock | 0 | 0 | 1
  SOC: CARDIAC DISORDERS, PT: Cardiomyopathy | 0 | 0 | 1
  SOC: ENDOCRINE DISORDERS, Total | 0 | 1 | 0
  SOC: ENDOCRINE DISORDERS, PT: Androgen deficiency | 0 | 1 | 0
  SOC: EYE DISORDERS, Total | 0 | 0 | 1
  SOC: EYE DISORDERS, PT: Lacrimation increased | 0 | 0 | 1
  SOC: GASTROINTESTINAL DISORDERS, Total | 3 | 15 | 3
  SOC: GASTROINTESTINAL DISORDERS, PT: Abdominal pain | 0 | 1 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Abdominal pain lower | 0 | 1 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Abdominal pain upper | 0 | 3 | 2
  SOC: GASTROINTESTINAL DISORDERS, PT: Constipation | 0 | 3 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Diarrhoea | 0 | 3 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Gastrooesophageal reflux disease | 0 | 1 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Inguinal hernia | 1 | 0 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Nausea | 2 | 8 | 3
  SOC: GASTROINTESTINAL DISORDERS, PT: Toothache | 1 | 0 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Vomiting | 2 | 13 | 3
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, Total | 2 | 11 | 1
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Chest pain | 0 | 0 | 1
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Fatigue | 1 | 6 | 0
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Infusion site reaction | 0 | 1 | 0
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Mass | 0 | 1 | 0
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Pyrexia | 1 | 8 | 0
  SOC: HEPATOBILIARY DISORDERS, Total | 0 | 2 | 1
  SOC: HEPATOBILIARY DISORDERS, PT: Liver injury | 0 | 2 | 1
  SOC: INFECTIONS AND INFESTATIONS, Total | 0 | 7 | 1
  SOC: INFECTIONS AND INFESTATIONS, PT: Cellulitis | 0 | 1 | 0
  SOC: INFECTIONS AND INFESTATIONS, PT: Conjunctivitis | 0 | 1 | 0
  SOC: INFECTIONS AND INFESTATIONS, PT: Influenza | 0 | 1 | 0
  SOC: INFECTIONS AND INFESTATIONS, PT: Molluscum contagiosum | 0 | 1 | 0
  SOC: INFECTIONS AND INFESTATIONS, PT: Nasopharyngitis | 0 | 2 | 0
  SOC: INFECTIONS AND INFESTATIONS, PT: Parainfluenzae virus infection | 0 | 0 | 1
  SOC: INFECTIONS AND INFESTATIONS, PT: Sinusitis | 0 | 3 | 0
  SOC: INFECTIONS AND INFESTATIONS, PT: Tooth abscess | 0 | 1 | 0
  SOC: INFECTIONS AND INFESTATIONS, PT: Urinary tract infection | 0 | 0 | 1
  SOC: INFECTIONS AND INFESTATIONS, PT: Viral upper respiratory tract infection | 0 | 1 | 0
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, Total | 0 | 6 | 1
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Contusion | 0 | 1 | 0
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Fall | 0 | 5 | 0
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Joint dislocation | 0 | 1 | 0
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Joint injury | 0 | 1 | 0
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Ligament sprain | 0 | 1 | 0
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Post procedural contusion | 0 | 1 | 0
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Procedural pain | 0 | 0 | 1
  SOC: INJURY, POISONING AND PROCEDURAL COMPLICATIONS, PT: Skin abrasion | 0 | 1 | 0
  SOC: INVESTIGATIONS, Total | 0 | 6 | 2
  SOC: INVESTIGATIONS, PT: Amylase increased | 0 | 1 | 0
  SOC: INVESTIGATIONS, PT: Complement factor C4 decreased | 0 | 5 | 0
  SOC: INVESTIGATIONS, PT: Cystatin C increased | 0 | 1 | 0
  SOC: INVESTIGATIONS, PT: Glutamate dehydrogenase increased | 0 | 3 | 0
  SOC: INVESTIGATIONS, PT: Hepatic enzyme increased | 0 | 0 | 1
  SOC: INVESTIGATIONS, PT: Lipase increased | 0 | 1 | 0
  SOC: INVESTIGATIONS, PT: Troponin increased | 0 | 0 | 1
  SOC: METABOLISM AND NUTRITION DISORDERS, Total | 2 | 8 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Decreased appetite | 2 | 6 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Dehydration | 0 | 5 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Hyperuricaemia | 0 | 1 | 0
  SOC: MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS, Total | 2 | 3 | 2
  SOC: MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS, PT: Arthralgia | 0 | 0 | 2
  SOC: MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS, PT: Back pain | 0 | 0 | 1
  SOC: MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS, PT: Myalgia | 0 | 1 | 0
  SOC: MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS, PT: Osteopenia | 1 | 0 | 0
  SOC: MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS, PT: Pain in extremity | 1 | 1 | 0
  SOC: NERVOUS SYSTEM DISORDERS, Total | 2 | 7 | 3
  SOC: NERVOUS SYSTEM DISORDERS, PT: Dizziness | 1 | 0 | 0
  SOC: NERVOUS SYSTEM DISORDERS, PT: Headache | 0 | 7 | 3
  SOC: NERVOUS SYSTEM DISORDERS, PT: Lethargy | 1 | 0 | 0
  SOC: NERVOUS SYSTEM DISORDERS, PT: Migraine | 0 | 1 | 0
  SOC: PSYCHIATRIC DISORDERS, Total | 2 | 3 | 0
  SOC: PSYCHIATRIC DISORDERS, PT: Abnormal behaviour | 0 | 1 | 0
  SOC: PSYCHIATRIC DISORDERS, PT: Affect lability | 1 | 1 | 0
  SOC: PSYCHIATRIC DISORDERS, PT: Anxiety | 0 | 1 | 0
  SOC: PSYCHIATRIC DISORDERS, PT: Irritability | 0 | 1 | 0
  SOC: PSYCHIATRIC DISORDERS, PT: Mood altered | 1 | 0 | 0
  SOC: PSYCHIATRIC DISORDERS, PT: Suicidal ideation | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, Total | 0 | 4 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Acute kidney injury | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Chronic kidney disease | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Glycosuria | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Haematuria | 0 | 2 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Ketonuria | 0 | 2 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Proteinuria | 0 | 2 | 0
  SOC: RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS, Total | 0 | 4 | 0
  SOC: RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS, PT: Cough | 0 | 2 | 0
  SOC: RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS, PT: Epistaxis | 0 | 1 | 0
  SOC: RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS, PT: Oropharyngeal pain | 0 | 1 | 0
  SOC: RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS, PT: Rhinorrhoea | 0 | 1 | 0
  SOC: SKIN AND SUBCUTANEOUS TISSUE DISORDERS, Total | 0 | 3 | 1
  SOC: SKIN AND SUBCUTANEOUS TISSUE DISORDERS, PT: Ecchymosis | 0 | 0 | 1
  SOC: SKIN AND SUBCUTANEOUS TISSUE DISORDERS, PT: Rash | 0 | 2 | 0
  SOC: SKIN AND SUBCUTANEOUS TISSUE DISORDERS, PT: Urticaria | 0 | 1 | 0
  SOC: VASCULAR DISORDERS, Total | 0 | 2 | 0
  SOC: VASCULAR DISORDERS, PT: Hypertension | 0 | 2 | 0

3. Primary Outcome: Number of Participants With Treatment-Related TEAEs for 1-Year Follow-Up
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Any AE that started following start of treatment of PF-06939926 was counted as a TEAE. An SAE was an untoward medical occurrence that resulted in death, was life-threatening (immediate risk of death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect, or was considered to be an important medical event. Severe AE=an event that prevents normal everyday activities. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Treatment-related AEs and SAEs were determined by the investigator.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  TEAEs | 3 | 15 | 3
  SAEs | 0 | 3 | 2
  Severe AEs | 0 | 2 | 2

4. Primary Outcome: Number of Participants With Treatment-Related TEAEs by SOC and PT for 1-Year Follow-Up
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Any AE that started following start of treatment of PF-06939926 was counted as a TEAE. For this outcome measure, TEAEs were reported according to MedDRA version 25.0 SOC and PT. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Treatment-related AEs were determined by the investigator.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, Total | 2 | 9 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Anaemia | 0 | 2 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Haemolysis | 0 | 1 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Haemolytic uraemic syndrome | 0 | 0 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Leukocytosis | 1 | 0 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Lymphopenia | 1 | 0 | 0
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Thrombocytopenia | 0 | 9 | 0
  SOC: CARDIAC DISORDERS, Total | 0 | 0 | 1
  SOC: CARDIAC DISORDERS, PT: Cardiogenic shock | 0 | 0 | 1
  SOC: GASTROINTESTINAL DISORDERS, Total | 2 | 15 | 3
  SOC: GASTROINTESTINAL DISORDERS, PT: Abdominal pain | 0 | 1 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Abdominal pain upper | 0 | 3 | 1
  SOC: GASTROINTESTINAL DISORDERS, PT: Diarrhoea | 0 | 1 | 0
  SOC: GASTROINTESTINAL DISORDERS, PT: Nausea | 2 | 8 | 3
  SOC: GASTROINTESTINAL DISORDERS, PT: Vomiting | 2 | 13 | 3
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, Total | 2 | 11 | 0
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Fatigue | 1 | 6 | 0
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Infusion site reaction | 0 | 1 | 0
  SOC: GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS, PT: Pyrexia | 1 | 8 | 0
  SOC: HEPATOBILIARY DISORDERS, Total | 0 | 2 | 1
  SOC: HEPATOBILIARY DISORDERS, PT: Liver injury | 0 | 2 | 1
  SOC: INVESTIGATIONS, Total | 0 | 6 | 2
  SOC: INVESTIGATIONS, PT: Amylase increased | 0 | 1 | 0
  SOC: INVESTIGATIONS, PT: Complement factor C4 decreased | 0 | 5 | 0
  SOC: INVESTIGATIONS, PT: Cystatin C increased | 0 | 1 | 0
  SOC: INVESTIGATIONS, PT: Glutamate dehydrogenase increased | 0 | 3 | 0
  SOC: INVESTIGATIONS, PT: Hepatic enzyme increased | 0 | 0 | 1
  SOC: INVESTIGATIONS, PT: Lipase increased | 0 | 1 | 0
  SOC: INVESTIGATIONS, PT: Troponin increased | 0 | 0 | 1
  SOC: METABOLISM AND NUTRITION DISORDERS, Total | 2 | 8 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Decreased appetite | 2 | 6 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Dehydration | 0 | 5 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Hyperuricaemia | 0 | 1 | 0
  SOC: NERVOUS SYSTEM DISORDERS, Total | 2 | 1 | 3
  SOC: NERVOUS SYSTEM DISORDERS, PT: Dizziness | 1 | 0 | 0
  SOC: NERVOUS SYSTEM DISORDERS, PT: Headache | 0 | 1 | 3
  SOC: NERVOUS SYSTEM DISORDERS, PT: Lethargy | 1 | 0 | 0
  SOC: RENAL AND URINARY DISORDERS, Total | 0 | 4 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Acute kidney injury | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Chronic kidney disease | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Glycosuria | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Haematuria | 0 | 2 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Ketonuria | 0 | 2 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Proteinuria | 0 | 2 | 0
  SOC: VASCULAR DISORDERS, Total | 0 | 2 | 0
  SOC: VASCULAR DISORDERS, PT: Hypertension | 0 | 2 | 0

5. Primary Outcome: Number of Participants With All-Causality SAEs by SOC and PT for 1-Year Follow-Up
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Any AE that started following start of treatment of PF-06939926 was counted as a TEAE. An SAE was an untoward medical occurrence that resulted in death, was life-threatening (immediate risk of death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect, or was considered to be an important medical event. For this outcome measure, TEAEs were reported according to MedDRA version 25.0 SOC and PT.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, Total | 0 | 1 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Haemolytic uraemic syndrome | 0 | 0 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Thrombocytopenia | 0 | 1 | 0
  SOC: CARDIAC DISORDERS, Total | 0 | 0 | 1
  SOC: CARDIAC DISORDERS, PT: Cardiogenic shock | 0 | 0 | 1
  SOC: INFECTIONS AND INFESTATIONS, Total | 0 | 0 | 1
  SOC: INFECTIONS AND INFESTATIONS, PT: Urinary tract infection | 0 | 0 | 1
  SOC: METABOLISM AND NUTRITION DISORDERS, Total | 0 | 1 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Dehydration | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, Total | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Acute kidney injury | 0 | 1 | 0

6. Primary Outcome: Number of Participants With Treatment-Related SAEs by SOC and PT for 1-Year Follow-Up
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Any AE that started following start of treatment of PF-06939926 was counted as a TEAE. An SAE was an untoward medical occurrence that resulted in death, was life-threatening (immediate risk of death), required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect, or was considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Treatment-related AEs and SAEs were determined by the investigator. For this outcome measure, TEAEs were reported according to MedDRA version 25.0 SOC and PT.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, Total | 0 | 1 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Haemolytic uraemic syndrome | 0 | 0 | 1
  SOC: BLOOD AND LYMPHATIC SYSTEM DISORDERS, PT: Thrombocytopenia | 0 | 1 | 0
  SOC: CARDIAC DISORDERS, Total | 0 | 0 | 1
  SOC: CARDIAC DISORDERS, PT: Cardiogenic shock | 0 | 0 | 1
  SOC: METABOLISM AND NUTRITION DISORDERS, Total | 0 | 1 | 0
  SOC: METABOLISM AND NUTRITION DISORDERS, PT: Dehydration | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, Total | 0 | 1 | 0
  SOC: RENAL AND URINARY DISORDERS, PT: Acute kidney injury | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality for 1-Year Follow-Up - Hematology
Description: Following hematologic parameters were analyzed for laboratory examination: hemoglobin, hematocrit, red blood cell (RBC) count, platelet count, white blood cell count, total neutrophils, absolute neutrophils (ANC), eosinophils, monocytes, basophils, lymphocytes, red blood cell indices, and haptoglobin. Laboratory abnormalities with occurrence in at least 1 participant are reported for this outcome measure. Baseline was defined as the last pre-dose measurement.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: Includes all enrolled participants who received PF-06939926. Participants were analyzed according to the intervention they actually received. Number of participants analyzed represents the total number of participants in each treatment group in the analysis population for this outcome measure. Number analyzed represents the number of participants who had reportable data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  Hemoglobin (g/dL) <0.8x Lower Limit of Normal (LLN) | 0 | 1 | 1
  Hematocrit (%)<0.8x LLN | 0 | 2 | 1
  Erythrocytes (10^6/mm3)<0.8x LLN | 0 | 1 | 1
  Platelets (10^3/mm3)<0.5x LLN | 0 | 5 | 1
  Erythrocyte Cell Morphology (No Unit)>0: number analyzed (Participants) | 2 | 14 | 3
  Erythrocyte Cell Morphology (No Unit)>0 | 0 | 1 | 1
  Leukocytes (10^3/mm3)>1.5x Upper Limit of Normal (ULN) | 0 | 2 | 1
  Lymphocytes (10^3/mm3)<0.8x LLN | 1 | 6 | 2
  Lymphocytes (10^3/mm3)>1.2x ULN | 0 | 2 | 1
  Lymphocytes Atypical (10^3/mm3)>0: number analyzed (Participants) | 1 | 9 | 2
  Lymphocytes Atypical (10^3/mm3)>0 | 1 | 9 | 2
  Neutrophils (10^3/mm3)<0.8x LLN | 0 | 2 | 0
  Neutrophils (10^3/mm3)>1.2x ULN | 1 | 7 | 2
  Neutrophils Band Form (10^3/mm3)>0.27: number analyzed (Participants) | 0 | 5 | 1
  Neutrophils Band Form (10^3/mm3)>0.27 |  | 0 | 1
  Basophils (10^3/mm3)>1.2x ULN | 0 | 1 | 0
  Eosinophils (10^3/mm3)>1.2x ULN | 1 | 2 | 0
  Monocytes (10^3/mm3)>1.2x ULN | 0 | 12 | 3
  Activated Partial Thromboplastin Time (sec)>1.1x ULN | 1 | 1 | 0
  Prothrombin Time (sec)>1.1x ULN | 1 | 7 | 2
  Neutrophils -TOTAL COUNT (10^3/mm3)<1.35 | 0 | 2 | 0
  Neutrophils -TOTAL COUNT (10^3/mm3)>8.15 | 2 | 14 | 2
  Myelocytes (10^3/mm3)>0: number analyzed (Participants) | 0 | 1 | 0
  Myelocytes (10^3/mm3)>0 |  | 1 |
  Haptoglobin (mg/dL)<30: number analyzed (Participants) | 0 | 13 | 3
  Haptoglobin (mg/dL)<30 |  | 3 | 1
  Haptoglobin (mg/dL)>200: number analyzed (Participants) | 0 | 13 | 3
  Haptoglobin (mg/dL)>200 | 0 | 10 | 3

8. Primary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality for 1-Year Follow-Up - Clinical Chemistry
Description: Following parameters for clinical chemistry were analyzed for laboratory examination: blood urea nitrogen (BUN) and creatinine, glucose, calcium, sodium, potassium, chloride, total CO2 (bicarbonate), aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin (direct and indirect bilirubin), alkaline phosphatase, uric acid, albumin, total protein, serum phosphorus, cystatin C, creatine kinase, creatine kinase myocardial b fraction (CK-MB), amylase, lipase, gamma-glutamyl transferase (GGT), C-reactive protein (CRP), and cardiac troponin I. Laboratory abnormalities with occurrence in at least 1 participant are reported for this outcome measure. Baseline was defined as the last pre-dose measurement.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  Bilirubin (mg/dL)>1.5x ULN | 0 | 0 | 1
  Direct Bilirubin (mg/dL)>1.5x ULN: number analyzed (Participants) | 3 | 16 | 2
  Direct Bilirubin (mg/dL)>1.5x ULN | 0 | 0 | 1
  Aspartate Aminotransferase (U/L)>3.0x ULN | 3 | 16 | 3
  Alanine Aminotransferase (U/L)>3.0x ULN | 3 | 16 | 3
  Gamma Glutamyl Transferase (U/L)>3.0x ULN | 0 | 1 | 1
  Protein (g/dL)<0.8x LLN | 0 | 2 | 0
  Albumin (g/dL)<0.8x LLN | 0 | 0 | 1
  Urea Nitrogen (mg/dL)>1.3x ULN | 0 | 1 | 1
  Creatinine (mg/dL)>1.3x ULN | 0 | 1 | 1
  Urate (mg/dL)>1.2x ULN | 0 | 6 | 0
  Sodium (mEq/L)<0.95x LLN | 0 | 1 | 2
  Potassium (mEq/L)<0.9x LLN | 0 | 1 | 1
  Calcium (mg/dL)<0.9x LLN | 0 | 0 | 1
  Phosphate (mg/dL)<0.8x LLN | 0 | 2 | 1
  Bicarbonate (mEq/L)<0.9x LLN | 0 | 2 | 2
  Bicarbonate (mEq/L)>1.1x ULN | 0 | 1 | 0
  Glucose (mg/dL)>1.5x ULN | 0 | 4 | 2
  Creatine Kinase (U/L)>2.0x ULN | 3 | 16 | 3
  Triacylglycerol Lipase (U/L)>1.5x ULN | 0 | 0 | 1
  C-Reactive Protein High Sens (mg/dL)>1.1x ULN | 0 | 3 | 2
  Cystatin C (mg/L)>1.2x ULN | 0 | 3 | 1
  Creatine Kinase MB (ug/L)>2.0x ULN: number analyzed (Participants) | 3 | 16 | 2
  Creatine Kinase MB (ug/L)>2.0x ULN | 3 | 16 | 2
  Glutamate Dehydrogenase (U/L)>1.0x ULN | 2 | 10 | 3
  Glutamate Dehydrogenase (U/L)>2.0x ULN | 0 | 5 | 2
  Glutamate Dehydrogenase (U/L)>3.0x ULN | 0 | 3 | 2
  Ferritin (ng/mL)<23.9: number analyzed (Participants) | 0 | 13 | 3
  Ferritin (ng/mL)<23.9 | 0 | 8 | 0
  Ferritin (ng/mL)>336.2: number analyzed (Participants) | 0 | 13 | 3
  Ferritin (ng/mL)>336.2 | 0 | 11 | 3

9. Primary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality for 1-Year Follow-Up - Urinalysis
Description: Following parameters for urinalysis were analyzed for laboratory examination: pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, and microscopy. Laboratory abnormalities with occurrence in at least 1 participant are reported for this outcome measure. Baseline was defined as the last pre-dose measurement.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  URINE Ketones (No Unit)>=1 | 0 | 7 | 3
  URINE Protein (Scalar)>=1 | 0 | 2 | 1
  URINE Hemoglobin (No Unit)>=1 | 0 | 4 | 1
  URINE Nitrite (No Unit)>=1 | 0 | 1 | 0
  URINE Erythrocytes (/high-powered field [HPF])>=20: number analyzed (Participants) | 1 | 6 | 3
  URINE Erythrocytes (/high-powered field [HPF])>=20 | 0 | 1 | 0
  URINE Leukocytes (/HPF)>=20: number analyzed (Participants) | 0 | 12 | 2
  URINE Leukocytes (/HPF)>=20 |  | 1 | 0
  Granular Casts (/low-power field [LPF])>1: number analyzed (Participants) | 0 | 1 | 0
  Granular Casts (/low-power field [LPF])>1 |  | 1 |
  Hyaline Casts (/LPF)>1: number analyzed (Participants) | 0 | 2 | 0
  Hyaline Casts (/LPF)>1 |  | 1 |
  Uric Acid Crystals (/LPF)>=0.5: number analyzed (Participants) | 0 | 2 | 0
  Uric Acid Crystals (/LPF)>=0.5 |  | 2 |
  Calcium Oxalate Crystals (/LPF)>=0.5: number analyzed (Participants) | 2 | 2 | 1
  Calcium Oxalate Crystals (/LPF)>=0.5 | 2 | 2 | 1
  Amorphous Crystals (/LPF)>=0.5: number analyzed (Participants) | 0 | 7 | 1
  Amorphous Crystals (/LPF)>=0.5 | 0 | 7 | 1
  Urine Microscopic Exam (Scalar)>=1: number analyzed (Participants) | 2 | 14 | 3
  Urine Microscopic Exam (Scalar)>=1 | 2 | 14 | 3

10. Primary Outcome: Change From Baseline on Left Ventricular Ejection Fraction as Measured by Cardiac Magnetic Resonance Imaging (MRI) for 1-Year Follow-Up
Description: Cardiac MRI was performed after thigh and upper limb MRI or on separate days within the required visit window. Change in LVEF is presented as percentages, and was calculated as [(stroke volume) / (end-diastolic volume)]*100%. Baseline is defined as the last pre-dose measurement. Change from baseline on Day 360 (ie, 1 year post dose) was reported for this outcome measure.
Time Frame: Baseline, 1 year post dose of PF-06839926 (Day 360)
Population: Includes all enrolled participants who received PF-06939926. Participants were analyzed according to the intervention they actually received. Number of participants analyzed represents the total number of participants in each treatment group in the analysis population and had reportable data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 14 | 2
Percentage | -0.7 (3.2) | -1.0 (4.3) | -3.1 (1.8)

11. Primary Outcome: Number of Participants With Electrocardiograms (ECGs) Meeting the Pre-Defined Categorical Criteria for 1-Year Follow-Up
Description: Triplicate ECG was performed after the participant had rested quietly for at least 10 minutes in a supine position. The pre-defined categorical criteria include PR interval aggregate (msec): value>=300, baseline>200 and percent change>=25%, baseline<=200 and percent change>=50%; QRS duration aggregate (msec): value>=140, percent change>=50%; QTcF interval aggregate (msec): 450<=value<480, 480<=value<500, value>=500, 30<=change<60, change>=60. Only the category(ies) with at least 1 participant meeting the pre-defined criterion is/are reported for this outcome measure. Baseline for ECG was defined as the measurement before the Day 1 study drug administration.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants | 1 | 2 | 0

12. Primary Outcome: Number of Participants With Positive Responses on Columbia-Suicide Severity Rating Scale (C-SSRS) According to the Columbia Classification Algorithm of Suicide Assessment (C-CASA) Categories
Description: C-SSRS is a participant rated questionnaire to assess whether participant experienced the following: completed suicide(1), suicide attempt(2)("Yes" on "actual attempt"), preparatory acts toward imminent suicidal behavior(3)("Yes" on "preparatory acts or behavior"), suicidal ideation(4)("Yes" on "wish to be dead","non-specific active suicidal thoughts","active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent), any suicidal behavior or ideation, self-injurious behavior(7)("Yes" on "Has subject engaged in non-suicidal self-injurious behavior"). Yes/No responses are mapped to C-CASA categories. C-SSRS was conducted with the participant's care giver/legal guardian on the participant's behalf throughout the study for participants<=12 years of age at screening. Baseline is defined as the last predose measurement. Number of participants with responses of "Yes" is reported for this outcome measure.
Time Frame: Baseline, Day 7, Day 14, Day 180, and Day 360
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  Baseline: Lifetime <1> Completed Suicide | 0 | 0 | 0
  Baseline: Lifetime <2> Suicide Attempt | 0 | 0 | 0
  Baseline: Lifetime <3> Preparatory Acts towards Imminent Suicidal Behavior | 0 | 0 | 0
  Baseline: Lifetime <4> Suicidal Ideation | 0 | 1 | 0
  Baseline: Lifetime <7> Self-injurious behavior, no suicidal intent | 0 | 0 | 0
  Baseline: Since Last Visit <1> Completed Suicide | 0 | 0 | 0
  Baseline: Since Last Visit <2> Suicide Attempt | 0 | 0 | 0
  Baseline: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior | 0 | 0 | 0
  Baseline: Since Last Visit <4> Suicidal Ideation | 0 | 0 | 0
  Baseline: Since Last Visit <7> Self-injurious behavior, no suicidal intent | 0 | 0 | 0
  Day 7: Since Last Visit <1> Completed Suicide: number analyzed (Participants) | 1 | 0 | 0
  Day 7: Since Last Visit <1> Completed Suicide | 0 | 0 | 0
  Day 7: Since Last Visit <2> Suicide Attempt: number analyzed (Participants) | 1 | 0 | 0
  Day 7: Since Last Visit <2> Suicide Attempt | 0 | 0 | 0
  Day 7: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior: number analyzed (Participants) | 1 | 0 | 0
  Day 7: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior | 0 | 0 | 0
  Day 7: Since Last Visit <4> Suicidal Ideation: number analyzed (Participants) | 1 | 0 | 0
  Day 7: Since Last Visit <4> Suicidal Ideation | 0 | 0 | 0
  Day 7: Since Last Visit <7> Self-injurious behavior, no suicidal intent: number analyzed (Participants) | 1 | 0 | 0
  Day 7: Since Last Visit <7> Self-injurious behavior, no suicidal intent | 0 | 0 | 0
  Day 14: Since Last Visit <1> Completed Suicide: number analyzed (Participants) | 0 | 13 | 2
  Day 14: Since Last Visit <1> Completed Suicide | 0 | 0 | 0
  Day 14: Since Last Visit <2> Suicide Attempt: number analyzed (Participants) | 0 | 13 | 2
  Day 14: Since Last Visit <2> Suicide Attempt | 0 | 0 | 0
  Day 14: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior: number analyzed (Participants) | 0 | 13 | 2
  Day 14: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior | 0 | 0 | 0
  Day 14: Since Last Visit <4> Suicidal Ideation: number analyzed (Participants) | 0 | 13 | 2
  Day 14: Since Last Visit <4> Suicidal Ideation | 0 | 0 | 0
  Day 14: Since Last Visit <7> Self-injurious behavior, no suicidal intent: number analyzed (Participants) | 0 | 13 | 2
  Day 14: Since Last Visit <7> Self-injurious behavior, no suicidal intent | 0 | 0 | 0
  Day 180: Since Last Visit <1> Completed Suicide: number analyzed (Participants) | 3 | 14 | 2
  Day 180: Since Last Visit <1> Completed Suicide | 0 | 0 | 0
  Day 180: Since Last Visit <2> Suicide Attempt: number analyzed (Participants) | 3 | 14 | 2
  Day 180: Since Last Visit <2> Suicide Attempt | 0 | 0 | 0
  Day 180: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior: number analyzed (Participants) | 3 | 14 | 2
  Day 180: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior | 0 | 0 | 0
  Day 180: Since Last Visit <4> Suicidal Ideation: number analyzed (Participants) | 3 | 14 | 2
  Day 180: Since Last Visit <4> Suicidal Ideation | 0 | 0 | 1
  Day 180: Since Last Visit <7> Self-injurious behavior, no suicidal intent: number analyzed (Participants) | 3 | 14 | 2
  Day 180: Since Last Visit <7> Self-injurious behavior, no suicidal intent | 0 | 0 | 0
  Day 360: Since Last Visit <1> Completed Suicide: number analyzed (Participants) | 3 | 16 | 2
  Day 360: Since Last Visit <1> Completed Suicide | 0 | 0 | 0
  Day 360: Since Last Visit <2> Suicide Attempt: number analyzed (Participants) | 3 | 16 | 2
  Day 360: Since Last Visit <2> Suicide Attempt | 0 | 0 | 0
  Day 360: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior: number analyzed (Participants) | 3 | 16 | 2
  Day 360: Since Last Visit <3> Preparatory Acts towards Imminent Suicidal Behavior | 0 | 0 | 0
  Day 360: Since Last Visit <4> Suicidal Ideation: number analyzed (Participants) | 3 | 16 | 2
  Day 360: Since Last Visit <4> Suicidal Ideation | 0 | 0 | 0
  Day 360: Since Last Visit <7> Self-injurious behavior, no suicidal intent: number analyzed (Participants) | 3 | 16 | 2
  Day 360: Since Last Visit <7> Self-injurious behavior, no suicidal intent | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Vital Signs Meeting the Pre-Defined Categorical Criteria for 1-Year Follow-Up
Description: Vital signs consisted of blood pressure, respiratory rate, and heart rate, was obtained with these measurements at the following timepoints: within 30 minutes before and approximately 30 minutes, 1, 2, 4, 8, and 24 hours after the start of the infusion, and on Days 4, 7, 10, 14, 30, 90, 180, and 360. Baseline was defined as the last pre-dose recording. Number of participants who had at least 1 vital sign measurement at the specified timepoints meeting the pre-defined criteria from baseline up to the end of 1-year follow-up is reported for this outcome measure.
Time Frame: Baseline up to 1 year post dose of PF-06939926
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
Number analyzed (Participants) | 3 | 16 | 3
Participants
  Respiratory Rate: value<14 breaths/min for aged 6-12 years: number analyzed (Participants) | 3 | 16 | 0
  Respiratory Rate: value<14 breaths/min for aged 6-12 years | 0 | 0 |
  Respiratory Rate: value>22 breaths/min for aged 6-12 years: number analyzed (Participants) | 3 | 16 | 0
  Respiratory Rate: value>22 breaths/min for aged 6-12 years | 3 | 16 |
  Respiratory Rate: value<12 breaths/min for aged 13-18 years: number analyzed (Participants) | 0 | 0 | 3
  Respiratory Rate: value<12 breaths/min for aged 13-18 years |  |  | 0
  Respiratory Rate: value>20 breaths/min for aged 13-18 years: number analyzed (Participants) | 0 | 0 | 3
  Respiratory Rate: value>20 breaths/min for aged 13-18 years |  |  | 3
  Supine Diastolic Blood Pressure: value<50 mmHg: number analyzed (Participants) | 3 | 16 | 2
  Supine Diastolic Blood Pressure: value<50 mmHg | 1 | 5 | 0
  Supine Diastolic Blood Pressure: increase>=20 mmHg: number analyzed (Participants) | 3 | 16 | 2
  Supine Diastolic Blood Pressure: increase>=20 mmHg | 0 | 2 | 0
  Supine Diastolic Blood Pressure: decrease>=20 mmHg: number analyzed (Participants) | 3 | 16 | 2
  Supine Diastolic Blood Pressure: decrease>=20 mmHg | 1 | 2 | 1
  Supine Heart Rate: value<40 beats per minute (bpm): number analyzed (Participants) | 3 | 16 | 2
  Supine Heart Rate: value<40 beats per minute (bpm) | 0 | 0 | 0
  Supine Heart Rate: value>120 bpm: number analyzed (Participants) | 3 | 16 | 2
  Supine Heart Rate: value>120 bpm | 0 | 1 | 1
  Supine Systolic Blood Pressure: value<70 mmHg + 2*age for aged 2-10 years: number analyzed (Participants) | 3 | 15 | 0
  Supine Systolic Blood Pressure: value<70 mmHg + 2*age for aged 2-10 years | 0 | 0 |
  Supine Systolic Blood Pressure: value<90 mmHg for aged 11 years and older: number analyzed (Participants) | 0 | 1 | 2
  Supine Systolic Blood Pressure: value<90 mmHg for aged 11 years and older |  | 1 | 0
  Supine Systolic Blood Pressure: increase from baseline>=30 mmHg: number analyzed (Participants) | 3 | 16 | 2
  Supine Systolic Blood Pressure: increase from baseline>=30 mmHg | 0 | 5 | 0
  Supine Systolic Blood Pressure: decrease from baseline>=30 mmHg: number analyzed (Participants) | 3 | 16 | 2
  Supine Systolic Blood Pressure: decrease from baseline>=30 mmHg | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to the end of 1-year follow-up (approximately 360 days)
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | PF-06939926: Low Dose, Ambulatory Cohort | PF-06939926: High Dose, Ambulatory Cohort | PF-06939926: High Dose, Non-Ambulatory Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/16 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 3/16 | 2/3
Other Adverse Events (participants affected / at risk) | 3/3 | 16/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06939926: Low Dose, Ambulatory Cohort (N=3) | PF-06939926: High Dose, Ambulatory Cohort (N=16) | PF-06939926: High Dose, Non-Ambulatory Cohort (N=3)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06939926: Low Dose, Ambulatory Cohort (N=3) | PF-06939926: High Dose, Ambulatory Cohort (N=16) | PF-06939926: High Dose, Non-Ambulatory Cohort (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 8 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Androgen deficiency (Endocrine disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 2
Constipation (Gastrointestinal disorders) | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 8 | 3
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 13 | 3
Chest pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 6 | 0
Infusion site reaction (General disorders) | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 8 | 0
Liver injury (Hepatobiliary disorders) | 0 | 2 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Molluscum contagiosum (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 3 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 5 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 1 | 0
Complement factor C4 decreased (Investigations) | 0 | 5 | 0
Cystatin C increased (Investigations) | 0 | 1 | 0
Glutamate dehydrogenase increased (Investigations) | 0 | 3 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 1 | 0
Troponin increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 7 | 3
Lethargy (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 1 | 0
Affect lability (Psychiatric disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2 | 0
Ketonuria (Renal and urinary disorders) | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/02/NCT03362502/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT03362502/SAP_001.pdf